CLINICAL TRIAL: NCT05840107
Title: CAR-T Injection in Transplant In-Eligible Newly Diagnosed Multiple Myeloma Patients
Brief Title: Study of FasT CAR-T GC012F Injection NDMM Patients
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Collaborators: Gracell Biotechnologies (Shanghai) Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Juan Du, Director of Hematology Department, Shanghai Changzheng Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC012F-322
Record Dates: First submitted 2023-04-22; First posted 2023-05-03 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GC012F treatment (Experimental): CAR-T will be infused at a dose of 0.6,1.5,3 x 10^5 CAR-T cells/kg after receiving lymphodepleting chemotherapy. Lenalidomide maintenance therapy will be given post month 6 at physicians' choice.
  Interventions: Biological: GC012F injection

INTERVENTIONS:
Biological: GC012F injection — GC012F injection is an autologous dual CAR-T targeted BCMA and CD19. A single infusion of CAR-T cells will be administered intravenously

SUMMARY:
This is a single-arm, single-center, open-label clinical study to evaluate the safety and efficacy of CAR-T in patients with NDMM.

DETAILED DESCRIPTION:
9-18 evaluable subjects are planned to be enrolled in this study. Apheresis will be carried out in subjects who meet eligible criteria, and total 2 cycles of induction therapy (three-drug combination regimen based on bortezomib with details determined by the investigator according to the patient's condition) will be selectively given to subjects before or after apheresis. Next, subjects will receive a single infusion of CAR-T, and the efficacy assessments will be performed at 1st month, 3rd months, and every 3 months within 2 years until the end of the trial (MRD testing is required for each efficacy assessment)

1.Efficacy assessments performed at the 1st month after infusion:

1. <PR: Protocol change or follow-up decided by the investigator.
2. ≥PR: Follow-up.

2.Efficacy assessments performed at the 3rd month after infusion and every 3 months thereafter:

1. <VGPR: Protocol change or follow-up decided by the investigator.
2. ≥VGPR: Maintenance treatment using lenalidomide until progress disease or clinical trial intolerance or termination of trial.

After signing the informed consent form (ICF), subjects will be followed up for efficacy and safety until 2 years after CAR-T infusion, or disease progression, or death, or withdrawal of consent, or any intolerable toxicity, whichever comes first. All AEs in subjects, especially infection related symptoms and signs, will be closely monitored during follow-up, and prophylactic treatment will be administered according to clinical practice when necessary. In case of disease progression within 2 years after CAR-T infusion, treatment will be administered according to clinical practice, and the survival follow-up (only for the survival status) will be performed every 12 weeks±14 days (2 weeks) until 2 years after infusion, or death, or withdrawal of consent, whichever comes first. For subjects who have undergone transportation or any other clinical routine treatments after CAR-T infusion, survival follow-up will be also performed as described above.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 when signing informed consent form（ICF）
2. Documented evidence of multiple myeloma at diagnosis as defined by IMWG guidelines ,monoclonal plasma cells in the bone marrow ≥10% and/or serum M protein ≥ 3 g/dL and/or 24h urine light chain ≥ 500 mg and/or presence of a biopsy proven plasmacytomas, not meet evidence of Smoldering Myeloma with SLiM/CRAB syptoms, and meet at least 2 of a-c or meet d of the following criteria at screening:

   1. Serum M protein ≥ 2 g/dL;
   2. Serum involved / uninvolved free light chain ratio ≥ 20;
   3. Bone marrow involved with monoclonal plasma cells ≥20% ;
   4. With Cytogenetic high-risk markers.
3. Or documented evidence of multiple myeloma at diagnosis as defined by IMWG guidelines CRAB (calcium elevation, renal insufficiency, anemia, and bone abnormalities)/SLiM criteria, monoclonal plasma cells in the bone marrow ≥10% or presence of a biopsy proven plasmacytomas, and measurable secretory disease according to IMWG criteria meet one or more of the following criteria at screening:

   1. Serum M protein ≥ 1 g/dL;
   2. Urine M protein ≥ 200 mg/24h;
   3. Serum free light chain sFLC ≥ 10 mg/dL with abnormal serum immunoglobulin κ/λ free light chain ratio.
4. ECOG score was 0-3 at screen;
5. Estimated life expectancy ≥3 months;
6. Absolute neutrophil count (ANC) ≥ 1.5×10^9/L without use of growth factors;
7. Platelet count ≥ 50×10^9/L without transfusion support within 7 days before the screen;
8. Hemoglobin≥ 60 g/L;
9. Adequate functional reserve of organs:

   1. ALT/AST ≤ 2.5× ULN(Upper Limit of Normal);
   2. Creatinine clearance ≥ 15mL/min;
   3. Serum total bilirubin ≤ 1.5×ULN, except in subjects with congenital bilirubinemia,then direct bilirubin ≤ 1.5×ULN;
   4. The left ventricular ejection fraction (LVEF)≥50%, and no clinically significant ECG abnormalities were found;
   5. Basic oxygen saturation in natural indoor air: SPO2>92%.
10. Adequate venous access for apheresis collection, and no other contraindications to apheresis;
11. Subjects and sexual partner with fertility are willing to use effective and reliable method of contraception for at least 1 year after CAR-T cell infusion, serum HCG should be negative in females with fertility both at screening and baseline;
12. Subjects must sign a written informed consent.

Exclusion Criteria:

1. Patients who are transplant eligible high-risk patients and plan to adopt auto/allo-transplantation
2. Subject has had radiation therapy within 14 days of screening;
3. Subjects has plasma cell leukemia or POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes);
4. Subjects has a diagnosis of primary amyloidosis, Waldenstroem's disease, monoclonal gammopathy of undetermined significance, or smoldering multiple myeloma;
5. Having other tumors (excluding non-melanoma skin cancer and cervical cancer in situ bladder cancer and breast cancer that have been disease-free for more than 5 years);
6. Evidence of serious mental disorders or changes in mental status, or the presence of central nervous system or diseases, such as seizures, cerebrovascular ischemia/hemorrhage, dementia, cerebellar diseases, or autoimmune diseases involving CNS;
7. History of hereditary diseases such as Fanconi anemia, Schrader syndrome, Costerman syndrome, or any other known bone marrow failure syndrome;
8. Clinically significant cardiac disease including: uncontrolled cardiac arrhythmia or clinically significant ECG abnormalities, grade III-IV heart failure or myocardial infarction cardiac angioplasty or stenting unstable angina or other clinically significant cardiac conditions within one year prior to enrollment;
9. Presence of any indwelling catheter or drainage tube (e.g., percutaneous nephrostomy catheter indwelling catheter bile drainage tube or pleural/peritoneal/pericardial catheter) The use of a dedicated central venous catheter is permitted;
10. Confirmed or suspected CNS involved;
11. A positive virological result for any of the following: HIV, HCV, HBsAg（If HBcAg positive, DNA copies must below the LOQ）, TPPA;
12. Other severe viral or bacterial infections or uncontrolled systemic fungal infections are present;
13. Severe allergic history or allergic constitution;
14. There is a history of an autoimmune disease (e.g., Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus) that has resulted in terminal organ damage or requires systemic immunosuppressive/disease modulating drugs in the past 2 years;
15. Presence of lung disease (such as pulmonary fibrosis);
16. Subjects has had major surgery within 2 weeks before screen or has not fully recovered from surgery, or has surgery planned during the time the subject is expected to participate in the study;
17. Poor compliance due to physiological, family, social, and geographical factors, etc., and inability to comply with the research program and follow-up plan;
18. Pregnant or lactating women;
19. Investigator assessment deemed to be ineligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AE) after CAR-T infusion | Up to 1 year after patients infused with CAR-T injection
  An assessment of severity grade will be made according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), with the exception of cytokine release syndrome (CRS), and immune effector cellassociated neurotoxicity syndrome (ICANS). CRS and ICANS should be evaluated according to the American Society for Transplantation and Cellular Therapy (ASTCT) consensus grading
Percentage of patients with complete response (CR) and stringent complete response (sCR) after infusion | Up to 2 years after patients infused with CAR-T injection
overall response rate (ORR) | Up to 2 years after patients infused with CAR-T injection
  ORR defined as proportion of patients achieving PR or better based on IMWG defined response criteria
Percentage of patients with minimal residual disease (MRD) negative in CR/sCR patients at landmark analysis | Up to 2 years after patients infused with CAR-T injection
  MRD negative rate
Progress free survival (PFS) | Up to 2 years after patients infused with GC01 2F injection
  PFS is defined as the time interval from the initiation of induction therapy until disease progression or death (for any reason).
Duration of response (DOR) after CAR-T infusion | Up to 2 years after patients infused with GC01 2F injection
  DOR is defined as the time interval from the first assessment of sCR, CR, VGPR or PR to the first assessment of PD or death from any cause after CAR T infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Du, MD, Principal Investigator — Shanghai Changzheng Hospital
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China